CLINICAL TRIAL: NCT00376493
Title: Prolonged Treatment for Infected Abortion After Hospital Discharge.
Acronym: APA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The rate of cure in both arms was higher than expected
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Ricardo Francalacci Savaris, Hospital de Clínicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APA 05-452
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2007-12

CONDITIONS: Septic Abortion
Keywords: Abortion; Infection; Antibiotics; Treatment; Pregnancy complications
MeSH Terms: conditions — Abortion, Septic; Infections; Pregnancy Complications | interventions — Metronidazole; Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Use of antibiotics after hospital discharge
  Interventions: Drug: metronidazole and doxycycline
- 2 (Placebo Comparator): Use of placebo
  Interventions: Drug: metronidazole and doxycycline

INTERVENTIONS:
Drug: metronidazole and doxycycline — use of metronidazole 500mg/day and doxycycline 200mg/day up to 10 days

SUMMARY:
Patients with infected abortion will be treated with dilatation and curettage, intravenous antibiotics. The purpose of this study is to verify if it is necessary to keep the use of oral antibiotics after hospital discharge.

DETAILED DESCRIPTION:
The use of 7-10 days of treatment for infected/septic abortion is not based on clinical trials. A recent evidence showed that endometritis post cesarean section needs no treatment after hospital discharge. The objective of this study is to verify if this finding also applies to infected abortions.

After in hospital treatment, the patients will be randomized to the traditional treatment (metronidazole and doxycycline) or to placebo until 10 days of treatment is completed. Active follow-up will be done every 2 days, and the patient will be reevaluated at the end of treatment.

Cure will be defined as the absence of fever, pain and bleeding. Failure of treatment will be considered as the need for hospitalization or additional antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* History of intrauterine manipulation with contaminated objects.
* Vaginal secretion with fetid odor
* Presence of pus flowing through the cervical uterine
* Presence of peritonitis
* Leucocytosis (> 14,000 leucocytes/mL)
* Vasodilatation, bounding pulse and paradoxically warm periphery with tachycardia (Heart rate> 110 bpm)
* Cyanosis and/or paleness
* tachypnea(> 30mpm)
* Arterial hypotension (SAP< 90mmHg)
* Oliguria
* Fever (> or = than 37,8°C)

Exclusion Criteria:

* Refusal to participate in the project
* Prior use of antibiotics within one week
* Known allergy to Doxycycline or Metronidazole
* Presence of tubo-ovarian abscess

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Hospital re-admission | 7 days after hospital discharge

SECONDARY OUTCOMES:
minimal or absent vaginal bleeding | 7 days after hospital discharge
walking normally | 7 days after hospital discharge
important decrease of pain | 7 days after hospital discharge
no fever | 7 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo F Savaris, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre; Adriani O Galão, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Stubblefield PG, Grimes DA. Septic abortion. N Engl J Med. 1994 Aug 4;331(5):310-4. doi: 10.1056/NEJM199408043310507. PMID 8022443
- [Background] Tamussino K. Postoperative infection. Clin Obstet Gynecol. 2002 Jun;45(2):562-73. doi: 10.1097/00003081-200206000-00026. No abstract available. PMID 12048413
- [Background] Turnquest MA, How HY, Cook CR, O'Rourke TP, Cureton AC, Spinnato JA, Brown HL. Chorioamnionitis: is continuation of antibiotic therapy necessary after cesarean section? Am J Obstet Gynecol. 1998 Nov;179(5):1261-6. doi: 10.1016/s0002-9378(98)70143-7. PMID 9822512
- [Background] Faro S. Postpartum endometritis. Clin Perinatol. 2005 Sep;32(3):803-14. doi: 10.1016/j.clp.2005.04.005. PMID 16085035
- [Background] French LM, Smaill FM. Antibiotic regimens for endometritis after delivery. Cochrane Database Syst Rev. 2004 Oct 18;(4):CD001067. doi: 10.1002/14651858.CD001067.pub2. PMID 15495005
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Hollis S, Campbell F. What is meant by intention to treat analysis? Survey of published randomised controlled trials. BMJ. 1999 Sep 11;319(7211):670-4. doi: 10.1136/bmj.319.7211.670. PMID 10480822